CLINICAL TRIAL: NCT06470594
Title: Superficial and Deep Endometriosis: Role of Systemic Inflammation as a Marker of Clinical, Surgical, and Reproductive Outcomes
Acronym: ESPRIMO-CCR
Status: Recruiting | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Gaetano Riemma, MD, University of Campania Luigi Vanvitelli
Other Study IDs: 0016489/i
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Superficial Endometriosis: Laparoscopic excision of superficial (peritoneal) endometriotic implants
- Ovarian Endometriosis: Laparoscopic excision of ovarian endometrioma/s
- Deep Infiltrating Endometriosis (DIE): Laparoscopic excision of DIE

SUMMARY:
Primary aim of this study is to evaluate the change in systemic inflammation parameters after surgery for superficial, ovarian or deep endometriosis. Secondary objectives focus on correlating these parameters to clinical outcomes, in patients with pelvic pain, and reproductive outcomes, in women desiring offspring.

Participants already scheduled for surgery as part of their endometriosis care will be followed regarding the abovementioned outcomes after calculation of pre and postsurgical systemic inflammation markers (neutrophil to lymphocyte ratio; platelet to lymphocyte ratio and lymphocyte to monocyte ratio)

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 45 years.
* Postoperative follow-up of at least 12 months;
* Signature of informed consent regarding laparoscopic surgical treatment.
* Signature of informed consent to the processing of personal data duly documented by medical records.

Exclusion Criteria:

* Failure to sign informed consent for laparoscopic surgical treatment
* Histologic diagnosis of borderline tumor and/or ovarian carcinoma and/or mucinous cystadenoma and/or germ cell tumor or other malignancy of the genital tract
* postoperative follow-up of less than 12 months;
* documented history of inflammatory, rheumatologic, or immunologic disease; and
* failure to provide informed consent for personal data processing.

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: Women with chronic pelvic pain and/or infertility with a sonographic or MRI ascertained suspicion of endometriosis.
Sampling Method: Probability Sample
Enrollment: 138 (Estimated)
Dates: Start 2024-05-29 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Neutrophil to lymphocyte ratio | Measured before and after (24 to 72 hours) surgery

SECONDARY OUTCOMES:
Platelet to lymphocyte ratio | Measured before and after (24 to 72 hours) surgery
Lymphocyte to monocyte ratio | Measured before and after (24 to 72 hours) surgery

CONTACTS AND LOCATIONS:
Locations (1):
- University of Campania Luigi Vanvitelli, Napoli, Italy